CLINICAL TRIAL: NCT03639584
Title: Investigating the Prevalence of Deficiency of Vitamin D in Critically Ill Patients and Its Effects on the Prognosis
Brief Title: Prevalence of Deficiency of Vitamin D in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805087RINB
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Vitamin D Deficiency; Critical Illness
Keywords: Vitamin D Deficiency; Critical Illness
MeSH Terms: conditions — Vitamin D Deficiency; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group 1: Patients admitted to ICU less than 48 hours and the anticipated stay is less than 5 days. Take blood sample on the day of enrollment.
- Group 2: Patients admitted to ICU less than 48 hours and the anticipated stay is longer than 5 days. Take blood sample on the day of enrollment, 7th, 14th, 21st, and 28th. Stop blood sample once exit.
- Group 3: Patients admitted to ICU 3~7 days. Take blood sample on the day of enrollment.
- Group 4: Patients admitted to ICU 8~14 days. Take blood sample on the day of enrollment.
- Group 5: Patients admitted to ICU 15~28 days. Take blood sample on the day of enrollment.

SUMMARY:
Vitamin D has been shown to related to clinical outcomes in critically ill patients. The object of this study is to investigate the prevalence of Vitamin D deficiency in critically ill patients with various length of ICU stay .

DETAILED DESCRIPTION:
Studies have revealed that the serum level of 25-hydroxyvitamin D, as known as calcidiol, is low in critically ill patients. The prevalence ranges from 26 to 82%. 25-hydroxyvitamin D deficiency is associated with longer ICU stay, higher medical cost and higher death rate in septic patients. 25-hydroxyvitamin D is a kind of hormone related to bone and mineral metabolism. Moreover, the receptors were found in almost all cells, and it is related to immune system, cytokine release, cellular proliferation and differentiation, angiogenesis, and muscular energy. The main source is skin metabolism triggered by sunshine and food consumption. It is subsequently converted to calcifediol in the liver and then calcitriol in the kidney (the active form). Its serum level is regulated by parathyroid hormone and serum calcium and phosphate. The critically ill patients are deprived of sunshine, suffered from poor nutrition support, impaired liver and kidney function, higher rate of consumption, and are under higher risk of deficiency. Nowadays, the studies about 25-hydroxyvitamin D in ICU patients were conducted mostly in Europe and America. There is no large-scale study in Taiwan or Asia. A randomized controlled study from Austria has shown large dose supply in patients with 25-hydroxyvitamin D deficiency could decrease the mortality.

The object of this multi-center study is to investigate the prevalence of 25-hydroxyvitamin D deficiency, the risk factors and the correlation with outcomes. The results could be a step-stone for future randomized controlled studies.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients

Exclusion Criteria:

* 1, Less than 20 years 2, BMI < 18 kg/m^2 3, Had large dose vit D within previous four weeks (over 3000 IU per day) 4, ICU admission within previous three months 5, Have disease affecting vit D level, calcium metabolism, bone metabolism such as parathyroid disease, Rickets, liver cirrhosis child C 6, Communication difficulty

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center, cross-sectional study involving four medical center in Taipei, Taiwan, which are National Taiwan University Hospital (NTUH), Far Eastern Memorial Hospital (FEMH), MacKay Memorial Hospital (MMH), and Taipei Medical University Hospital (TMUH). The target population is all the ICU patients, divided into four groups according to the length of ICU stay. The serum level of vit D, ICU event such as infection, ventilator dependency is to be recorded.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The prevalence of Vitamin D deficiency | 1 day at enrollment
  Investigate the prevalence of vitamin D deficiency among groups

SECONDARY OUTCOMES:
Difference of mortality on 28th and 90th day in group 2 | 90 days
  Compare the mortality of 28th and 90th day of patients with vitamin D deficiency and patients without vitamin D deficiency in group 2
Difference of mortality on 28th and 90th day in group 3, 4, and 5 | 90 days
  Compare the mortality of 28th and 90th day of patients with vitamin D deficiency and patients without vitamin D deficiency in group 3, 4, and 5
Serial changes of serum vitamin D levels in group 2 | 28 days
  investigate the serum vitamin D levels at different time points in group 2
Difference of 28-day ventialtor-free days | 28 days
  Compare the 28-day ventialtor-free days of patients with vitamin D deficiency and patients without vitamin D deficiency for all groups
Difference of 28-day ICU-free days | 28 days
  Compare the 28-day ICU-free days of patients with vitamin D deficiency and patients without vitamin D deficiency for all groups

CONTACTS AND LOCATIONS:
Overall Officials: Chung-Wei Chen, MD, Principal Investigator — Far Eastern Memorial Hospital; Li-Kuo Kuo, MD, Principal Investigator — Mackay Memorial Hospital; Kuo-Ching Yuan, MD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Kuo YT, Kuo LK, Chen CW, Yuan KC, Fu CH, Chiu CT, Yeh YC, Liu JH, Shih MC. Score-based prediction model for severe vitamin D deficiency in patients with critical illness: development and validation. Crit Care. 2022 Dec 21;26(1):394. doi: 10.1186/s13054-022-04274-9. PMID 36544226